CLINICAL TRIAL: NCT06269198
Title: Postoperative Complications in Cancer Patients Monitored With Intelligent Continuous Monitoring System Versus Standard of Care - a Randomized Clinical Trial
Brief Title: Postoperative Complications in Cancer Patients Monitored With Intelligent Continuous Monitoring System
Acronym: WARD-SX-RCT-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Bispebjerg Hospital (Other); Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Jesper Mølgaard, MD, PhD, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WARD - SX - RCT II
Record Dates: First submitted 2024-02-06; First posted 2024-02-21 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Complications; Cancer, Treatment-Related
Keywords: vital signs; continuous monitoring; wireless monitoring; postoperative physiology; postoperative complications
MeSH Terms: conditions — Postoperative Complications; Neoplasms, Second Primary

STUDY DESIGN:
Intervention Model Description: Randomisation stratified by study site
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be given information on group allocation. Care-providers will not be blinded, due to having to carry out the intervention.
  Investigator will not be blinded to carrie out roles such as safety surveillance, error-solving and quality assurance.
  Outcome assessor will be blinded to study allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Blinded data collection by the WARD-CSS without vital signs and active alerts displayed to the ward staff
- Intervention arm (Experimental): Monitoring by the WARD-CSS including vital signs and active alerts relayed to the nurses' smartphones during hospitalization
  Interventions: Device: WARD-CSS

INTERVENTIONS:
Device: WARD-CSS — Patients' continuously monitored vital signs will be recorded via a bedside tablet device (data not visible).
  The clinical staff will have access to the continuously monitored vital signs through a mobile device (smart phone) with a purpose-built app-based GUI displaying vital sign status and summaries, alarms, and device connectivity. The GUI will alert the clinical staff (acoustic and visual signals) when any of the predefined thresholds for deviating vital signs are exceeded.
  Other Names: Continuous vital signs monitoring with real-time alerts
  Arms: Intervention arm

SUMMARY:
The primary objective of this study is to determine the effect on complication severity of using a clinical monitoring system with automatic vital sign alerts in addition to routine monitoring versus routine monitoring alone in high-risk postoperative cancer patients within 30 days after surgery.

Other objectives include documentation of the severity of complications within seven days of surgery, frequency of serious adverse events, mortality, length of stay and delay of planned chemotherapy.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the effect on complication severity of using the WARD-CSS with automatic alerts in addition to routine monitoring versus routine monitoring alone in high-risk postoperative cancer patients within 30 days after surgery.

This study is a multicenter randomized controlled trial (RCT). Patients are randomly assigned to one of two parallel monitoring groups: (1)Intervention group - Monitoring by the WARD-CSS including vital signs and active alerts relayed to the nurses' smartphones during hospitalization. (2)Control group - Blinded data collection by the WARD-CSS without vital signs and active alerts displayed to the ward staff.

Both groups will receive routine vital signs monitoring (i.e. manual spot-checks) using the regional EWS/TOKS system according to current standards of care at the participating hospitals in the Capital Region or the Central Denmark Region.

The study is a collaboration between Rigshospitalet, Bispebjerg and Frederiksberg Hospital, and Hvidovre Hospital.

Patients will be recruited from abdominal (gastrointestinal, gynecological, or urological) surgery wards at the study sites.

Patients will be randomized post-surgery at the postoperative units/ post-anesthesia-care unit or after arrival at the ward. Continuous wireless monitoring (i.e., unblinded with alerts or blinded) will commence immediately after randomization in the study.

Only randomized patients will be included in the study population. Drop-outs prior to randomization will not be part of the study population.

The first 14 days of active enrollment at each new study site that has not previously used WARD-CSS will be used to align study procedures, verify system connectivity, etc. During this period, up to ten patients at each study site will be enrolled to be monitored similar to the intervention group. These run-in patients will not be randomized and will not be considered part of the study population.

ELIGIBILITY:
Inclusion Criteria:

* Admission for elective major abdominal (gastrointestinal, gynecological, or urological) surgery with the primary aim of radical surgery/removing suspected cancer tissue.
* At least two expected postoperative admission days
* Laparotomy or laparoscopy procedure estimated to last more than 2 hours.
* Co-enrolment of patients in other studies is acceptable but in studies involving interventions which potentially will affect the continuous monitoring of vital signs and/or the primary or secondary outcomes, an assessment of whether these patients can be co-enrolled in the WARD-RCT should be conferred with the WARD RCT steering committee.

Exclusion Criteria:

* Patient expected not to cooperate with study procedures
* Allergy to study materials (silicone, plaster)
* Impaired cognitive function (in uncertain cases assessed by a Mini Mental State Examination score < 24). (Protocol Appendix E)
* Patients with a pacemaker or Implantable Cardioverter Defibrillator (ICD) device
* Inability to give informed consent
* Patients with planned hyperthermic intraperitoneal chemotherapy (HIPEC) procedure or two-stage resections (two-stage hepatectomy, two-stage resection of malignant colorectal obstructions, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Overall complication severity - 30 days | 30 days after surgery
  Severity of complications assessed by the Comprehensive Complication Index (CCI) score. Complications are defined according to internationally agreed definitions of complications.
  CCI can take on numerical values in the scale from 0 (no complications) to 100 (patient deceased).

SECONDARY OUTCOMES:
Overall complication severity - 7 days | 7 days after surgery
  Severity of complications assessed by the Comprehensive Complication Index (CCI) score. Complications are defined according to internationally agreed definitions of complications.
  CCI can take on numerical values in the scale from 0 (no complications) to 100 (patient deceased).
Frequency of Serious adverse events | 30 days after surgery
  Frequency of Serious adverse events (SAE) SAE is defined by ICH-GCP criteria as: Any unfavourable medical occurrence that
  * results in death
  * is life-threatening
  * requires inpatient hospitalisation or prolongation of existing hospitalisation
  * results in persistent or significant disability/incapacity
  * is a congenital anomaly/birth defect
Days alive and out of hospital | 30 days after surgery
  Number of days alive and out of hospital
Days alive and out of hospital | 6 months after surgery
  Number of days alive and out of hospital
Time to initiation of post-operative adjuvant chemotherapy | Outcomes will be collected up to 2 year after surgery
  For patients scheduled to recieve postoperative chemotherapy, this is the time from surgery to initiation of post-operative adjuvant chemotherapy
Completion of post-operative adjuvant chemotherapy | Outcomes will be collected up to 2 year after surgery
  For patients scheduled to recieve postoperative chemotherapy, this is the number of patients that complete their post-operative adjuvant chemotherapy.

OTHER OUTCOMES:
Frequency of severe clinical complications | 30 days after surgery
  Frequency of severe clinical complications Defined as any complication fulfilling the Clavien-Dindo classification ≥2
ICU admission | 30 days after surgery.
  Number of patients with unplanned admission to the intensive care unit after surgery
Surgical reintervention of any kind | 30 days after primary-surgery
  Any unplanned surgical reintervention of any kind.
Post-discharge readmission | 6 months after surgery.
  Re-admission for any reason related to the operation or their respective cancer
Health-economic cost-effectiveness. | 2 years after surgery.
  Health-economic cost-effectiveness. Data will be collected from all available health care databases in the danish public health care system (ie. use of general practitioners, hospital admissions, hospital registered costs and services, work-leave periods) for a maximum follow up period of 2 years after primary surgery and analyzed when full datasets are available

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Mølgaard, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (3):
- Denmark (3):
  - Copenhagen University hospital - Rigshospitalet, Copenhagen, Other (Non US)
  - Bispebjerg Hospital, Copenhagen, Other (Non US)
  - Hvidovre Hospital, Hvidovre, Other (Non US)

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD